CLINICAL TRIAL: NCT03366389
Title: Evaluation of the Serum Levels of Apelin, Chemerin and Adiponectin Adipokines in Patients With Irritable Bowel Syndrome and Healthy Subjects
Brief Title: Serum Levels of Apelin, Chemerin and Adiponectin Adipokines in Irritable Bowel Syndrome and Healthy Subjects
Status: Completed | Type: Observational
Sponsor: Amir Abbasnezhad (Other)
Collaborators: Lorestan University of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Amir Abbasnezhad, Assistant Professor of Nutrition Science, Lorestan University of Medical Sciences
Organization: Lorestan University of Medical Sciences (Other)
Other Study IDs: Lums.REC.1396.266
Record Dates: First submitted 2017-11-10; First posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: patients with irritable bowel syndrome
- Control: Healthy subjects without any gastrointestinal disorders, chronic diseases and malignancy.

SUMMARY:
In this observational case-control study investigators aimed to assess the serum levels of adipokines such as Apelin, Chemerin and adiponectin in patients with irritable bowel syndrome (IBS), and compare it with healthy controls. Furthermore, investigators evaluated the possible correlation of these adipokines with IBS-QoL, IBSSS, GI symptoms and other clinical and psychological disorders.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18, and 80 years.
* IBS patients diagnosed according to the Rome III Diagnostic Criteria for Functional GI Disorders.

Exclusion Criteria:

* Any evidence of abdominal surgery or radiation
* celiac disease, or other primary GI illnesses
* GI infection obscuring IBS symptoms,
* using total parenteral nutrition therapy in the last 6 months
* pregnancy and lactation
* alcohol consumption
* concurrent chronic diseases such as diabetes, renal failure
* diagnosed and/or treated malignancy in the past 5 years
* anti-inflammatory drugs usage
* intake of vitamin D, omega-3, vitamin E, and calcium supplements
* being on a special diet or medication regimen during the last 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients were recruited from the outpatient clinic at the Lorestan University of Medical Sciences, Khorramabad, Iran, by an attendant gastroenterologist.
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2017-09-16 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
Serum levels of Apelin, Chemerin and adiponectin | in recruitment

SECONDARY OUTCOMES:
IBS-Quality of life (IBS-QoL) | in recruitment
  The Quality of life was assessed at the baseline and at the end of the study using a self-report QoL measure specific to IBS (IBS-QoL) with 34 items
IBS severity score system (IBSSS) | in recruitment
  Irritable bowel syndrome severity score system is validated for use in IBS patients, which included five clinically relevant items during a 10-day period: (i) severity of abdominal pain, (ii) frequency of abdominal pain, (iii) severity of abdominal distention or tightness, (iv) dissatisfaction with bowel habits, and (v) interference of IBS with life in general. Each item was scored on a scale from 0 to 100, and the sum of these five items was the score of IBS severity (range 0-500). Scores of 75-175, 175-300, and >300 indicated mild, moderate, and severe cases, respectively.
Gastrointestinal symptoms | in recruitment
Somatic Symptom | in recruitment
Personality | in recruitment
  Big Five Inventory Questionnaire
Perceived Stress Scale | in recruitment
  The Perceived Stress Scale (PSS) is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful.Higher PSS scores were associated with a greater vulnerability to stressful life-event-elicited depressive symptoms.
  PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. A short 4 item scale can be made from questions 2, 4, 5 and 10 of the PSS 10 item scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Lorestan university of medical sciences, Khorramabad, Iran

IPD SHARING:
Plan to Share IPD: Undecided